CLINICAL TRIAL: NCT04085705
Title: The Prevalence of Contact Allergies for Wound Dressings In Patients With Diabetic Foot Ulcers
Brief Title: The Prevalence of Contact Allergies for Wound Dressings In Patients With Diabetic Foot Ulcers (PAID Study)
Acronym: PAID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Visch MD, Principal Investigaor, Rijnstate Hospital
Other Study IDs: PAID study
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot; Contact Allergy
Keywords: Wound Dressing
MeSH Terms: conditions — Diabetic Foot; Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetic foot ulcers: All patients with diabetic foot ulcers will undergo a PATCH test to determine the prevalence of contact allergies against wound dressings.
  Interventions: Diagnostic Test: PATCH test

INTERVENTIONS:
Diagnostic Test: PATCH test — The PATCH test is a method used to determine whether a specific substance causes allergic inflammation of a patient's skin, in this case contact allergy for wound dressings. Two days after PATCH test is applied, the patches are removed. The next day, the presence of a contact allergy is determined.

SUMMARY:
Rationale: Foot ulcers among diabetics are common. The presence of a contact allergy limits the healing process. Contact allergies for wound dressings are common among patients with ulcers caused by venous insufficiency but less is known about contact allergies in diabetic patients with ulcers.

Objective: To determine the prevalence of contact allergies for wound dressings in patients with diabetic foot ulcers.

Study design: A prospective multicenter study.

Study population: Patients (n=139) with diabetic foot ulcers caused by type 1 or 2 diabetes mellitus treated at Rijnstate Hospital Arnhem, the Netherlands.

Main study parameters/endpoints: The primary study parameter is the presence of contact allergies for wound dressings.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: An allergy test is standard procedure at Rijnstate Hospital, there is no direct technique-related burden or risk for the patient. In addition, wound dressings can be adjusted in patients where a contact allergy is determined which will benefit the prognosis of these patients. The data of this study will give insight in the prevalence of contact allergies for wound dressings in patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
Foot ulcers among diabetics are common. In 2015, around 20,000 patients in the Netherlands had a diabetic foot ulcer.1 A study using data from Dutch general practices found a prevalence rate of 0.50% and a 4-year prevalence rate of 2.85%.2 For Europe, Zhang et al. estimated a pooled prevalence of 5.1% (95%CI: 4.1-6.0%).3 Prevalence rates increase with age.

The underlying mechanism of diabetic foot ulcers is most often solely neuropathy (60 to 70%), 15 to 20% have peripheral artery disease (PAD) only, and 15 to 20% have a mixture of both.4 Diabetic foot is more prevalent in males and more prevalent in type 2 diabetes than in type 1 diabetes3. Ulcers in patients without diabetes are mostly caused by venous insufficiency.5

Ulcers have a slow healing tendency. Around 15 percent of diabetic patients with an ulcer eventually have to amputate (a part of) the leg.1 Good wound care is therefore important. However, wound care can be delayed in the presence of a contact allergy. Contact allergy (synonym for contact sensitivity) is defined as an altered immune status of an individual induced by a particular sensitizing substance, a contact allergen. An individual in whom contact allergy has been induced will develop a secondary immune response if there is skin exposure to the same (or cross-reacting) allergen. This process is called elicitation, and will manifest as allergic contact dermatitis (type IV hypersensitivity).6 Allergic contact dermatitis, also termed allergic contact eczema, is defined as an inflammatory skin reaction caused by direct contact with noxious agents in the environment as a result of contact allergy.

Among patients with venous leg ulcers contact allergies is seen in around 50 percent of which 10-20% for wound dressings.7-10 The prevalence of contact allergies is getting higher and also increasing with the duration of the ulcer. 8,10 Wound dressings can cause allergic contact eczema (allergic contact dermatitis).

At present, the prevalence of contact allergies for wound dressings in diabetic patients with foot ulcers is unknown. With this study we want to gain insight in the prevalence of contact allergies in patients with diabetic foot ulcers and investigate if the prevalence of contact allergies among diabetic patients is as high as the prevalence in patients with venous leg ulcers.

Objective of the study:

The primary objective of this study is to determine the prevalence of contact allergies in patients with diabetic foot ulcers.

Study design:

This is a prospective, multi-centre study.

Study population:

The study population are high risk diabetic patients with a foot ulcer visiting the multidisciplinary consultation hour for diabetics at the clinic.

Diabetic patients are patients diagnosed with type 1 or type 2 diabetes.

Primary study parameters/outcome of the study:

The presence of contact allergy for wound dressings

Secundary study parameters/outcome of the study (if applicable):

The following factors will be gathered at baseline:

* Age
* Gender
* Diabetes type
* Duration of diabetes
* Medication use
* Ulcer characteristics like type, size, duration, progress (TEXAS classification)
* Number of past foot ulcers
* Duration of past foot ulcers
* Known allergies or atopy constitution
* Presence of allergic contact dermatitis around the wound
* Doses corticosteroid or antihistaminic therapy (not during PATCH testing)
* History of eczema

Parameters to define if there are other mechanisms besides diabetics underlying the ulcer:

* Ankle brachial index , toe pressure measurement or Transcutaneous oxygen pressure (TcPo2)
* Venous insufficiency which is measured by a venous duplex, if applicable

Parameters related with contact allergy or parameters that can influence the development of a contact allergy:

* Known allergy. If yes, which allergy/allergies?
* Duration of current ulcus cruris
* Number of past ulcers
* Treatment with wound dressing(s) current episode:

  * Duration of ulcer
* Treatment with wound dressing(s) prior episode(s)
* Prevalence of allergic contact dermatitis

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

Not applicable

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older;
* Diagnosed with type 1 or 2 diabetes mellitus;
* Diagnosed with diabetic foot ulcer;
* Provided written informed consent.

Exclusion Criteria:

* Patient unwilling or unlikely to comply with the study procedures
* Patient receiving systemic corticosteroid therapy during PATCH testing (patient should stop with corticosteroid therapy three days before PATCH testing, and may start when testing and reading is done)
* Patient receiving antihistaminic therapy during PATCH testing (patient should stop with antihistaminic therapy three days before PATCH testing, and may start when testing and reading is done)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are high risk diabetic patients with a foot ulcer visiting the multidisciplinary consultation hour for diabetics at the clinic.
  Diabetic patients are patients diagnosed with type 1 or type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Presence of contact allergy for wound dressings | 3 days after application of PATCH test
  The presence of contact allergy for wound dressings

SECONDARY OUTCOMES:
Presence of eczema | Collected at baseline
  Presence of eczema/dermatitis

OTHER OUTCOMES:
Ulcer duration | Collected at baseline
  Duration of ulcers
Past ulcers | Collected at baseline
  The number of ulcers in the past

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Visch, MD, Principal Investigator — Rijnstate
Locations (1):
- Rijnstate, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] Visch BM, Veen DV, Smeets L, Toeter R, Bon AV, Romijn D. The Prevalence of Contact Allergies for Wound Dressings in Patients With Diabetic Foot Ulcers (PAID Study), an Observational Prospective Trial. Int J Low Extrem Wounds. 2025 Apr 10:15347346251332028. doi: 10.1177/15347346251332028. Online ahead of print. PMID 40208179